CLINICAL TRIAL: NCT06498739
Title: Comparing the Perioperative Analgesic Effect of Two Different Volumes of Local Anesthetic Solution in Erector Spinae Plane Block in Patients Undergoing Modified Radical Mastectomy. A Randomized Comparative Study
Brief Title: Perioperative Analgesic Effect of Two Different Volumes of Local Anesthetic Solution in Erector Spinae Plane Block in Patients Undergoing Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmina Sayed, Assistant lecturer of anesthesiology and surgical ICU and pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MS-520-2022
Record Dates: First submitted 2023-12-13; First posted 2024-07-12 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Erector Spinae Plane Block; Modified Radical Mastectomy
MeSH Terms: interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane block (high concentration-low volume) (Other): Patients will preoperatively receive high concentration-low volume ultrasound guided Erector Spinae Plane block, and then the patient will be transferred to the operating room (one syringe of 15 ml bupivacaine 0.5% {15 ml bupivacaine 0.5% }, for each patient).
  Interventions: Drug: Erector spinae plane block(15 ml bupivacaine 0.5%)
- Erector Spinae Plane block (low concentration-high volume) (Other): Patients will preoperatively receive low concentration-high volume ultrasound guided Erector Spinae Plane block, and then the patient will be transferred to the operating room ) one syringe of 30ml bupivacaine 0.25% {15 ml bupivacaine 0.5% and 15ml normal saline}, for each patient.
  Interventions: Drug: Erector spinae plane block (15 ml bupivacaine 0.5% and 15ml normal saline)

INTERVENTIONS:
Drug: Erector spinae plane block(15 ml bupivacaine 0.5%) — Patients will preoperatively receive high concentration-low volume ultrasound guided Erector Spinae Plane block, and then the patient will be transferred to the operating room (one syringe of 15 ml bupivacaine 0.5% {15 ml bupivacaine 0.5% }, for each patient).
  Arms: Erector Spinae Plane block (high concentration-low volume)
Drug: Erector spinae plane block (15 ml bupivacaine 0.5% and 15ml normal saline) — Patients will preoperatively receive low concentration-high volume ultrasound guided Erector Spinae Plane block, and then the patient will be transferred to the operating room ) one syringe of 30ml bupivacaine 0.25% {15 ml bupivacaine 0.5% and 15ml normal saline}, for each patient.
  Arms: Erector Spinae Plane block (low concentration-high volume)

SUMMARY:
Comparing the perioperative analgesic effect of two different volumes of local anesthetic solution in erector spinae plane block in patients undergoing modified radical mastectomy. A randomized comparative study.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy among females with incidence of about 2.1 million women each year. Modified Radical Mastectomy (MRM) is one of the main surgical treatments of breast cancer.

Pain can be severe enough to cause long-term disabilities and interfere with sleep and performance of daily activities . Multiple regional techniques have been developed in recent years for postoperative analgesia of breast surgery inkling erector spinae plane block (ESPB) aiming to be effective and associated with less complications when compared to the gold standard techniques (thoracic epidural analgesia or paravertebral block). Ultrasound guided erector spinae plane block (ESPB) was described in 2016 as a novel regional anesthetic technique for acute and chronic thoracic pain, it has been used as a regional anesthetic technique for breast surgery based on case reports and case series. It is a paraspinal fascial plane block that involves injection of local anesthetic deep in the erector spinae muscle and superficial to the tips of the thoracic transverse processes. The site of injection is distant from the pleura, major blood vessels, and spinal cord.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 60 years.
* Genders eligible for study: female sex.
* American Society of Anesthesiologists (ASA) I-II.
* Undergoing modified radical mastectomy.
* Body mass index (BMI) from 18.5 to 30 kg.

Exclusion Criteria:

* Patient refusal.
* Known allergy to local anesthetics .
* Bleeding disorders; platelets count <50,000 ,prothrombin concentration < 60% or any coagulopathy disorder.
* Use of any anti-coagulants .
* Inability to provide informed consent.
* Neurological disorders.
* Patient with psychiatric disorders.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women undergoing modified radical mastectomy
Enrollment: 52 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperative
  Rescue analgesia will be provided in the form of intravenous morphine 3 mg boluses if the patient indicates visual analogue scale ≥ 4. The total amount of morphine given in 24 hours will be recorded for the two groups. A maximum dose of 0.5 mg/kg/24hours of morphine is allowed.
  Visual Analogue Scale (VAS) (0 represents "no pain" while 10 represents "the worst pain imaginable").

SECONDARY OUTCOMES:
Time 1st rescue analgesia | 24 hours postoperative
  All patients will receive paracetamol 1gm and intravenous ketorolac 30mg will be provided as a part of multimodal analgesia. Rescue analgesia will be provided in the form of intravenous morphine 3 mg boluses if the patient indicates visual analogue scale ≥ 4. The total amount of morphine given in 24 hours will be recorded for the two groups. A maximum dose of 0.5 mg/kg/24hours of morphine is allowed.
  Visual Analogue Scale (VAS) (0 represents "no pain" while 10 represents "the worst pain imaginable").
Pain score | 24 hours postoperative
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable").it will be assess at 0 , 4, 8, 12, 16, 20 and 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Univesity, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.